CLINICAL TRIAL: NCT03220386
Title: Methicillin-sensitive and Methicillin-resistant Staphylococcus Aureus (MSSA/MRSA) - Point-of-care-testing (POCT) in Clinical Decision Making
Acronym: EPICS-6
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Martin Moeckel, Professor Dr. med., Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EA1/055/17
Record Dates: First submitted 2017-05-08; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Staphylococcus Aureus
Keywords: staphylococcus aureus; nosocomial infection; decolonization; emergency department
MeSH Terms: conditions — Staphylococcal Infections; Cross Infection; Emergencies

STUDY DESIGN:
Intervention Model Description: Patients screened positive for nasal MSSA or MRSA colonization during their treatment in the emergency department receive a standardized decolonization Treatment (Octinidin nasal ointment and skin washing)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emergency Department patients (Other): All patients will be tested for nasal MSSA/MRSA-colonization. Patients tested positive for nasal MSSA/MRSA-colonization receive a decolonization treatment. This treatment includes octinidin nasal treatment and skin washings.
  Interventions: Other: Decolonization by nasal Octinidin treatment and skin washings

INTERVENTIONS:
Other: Decolonization by nasal Octinidin treatment and skin washings — Patients receive nasal Octinidin treatment and skin washings for five consecutive days

SUMMARY:
The study EPICS-6 consists of three study phases. Emergency Department patients are screened for nasal and pharyngeal colonisation with Methicillin sensitive and Methicillin resistant Staphylococcus aureus (MSSA/MRSA) using a point-of-care (POC)-PCR-testing method (cobas®LIAT®-System, Roche Molecular Systems Inc.) The first aim of this study is to describe the prevalence of MSSA/MRSA-colonisation in a routine cohort of Emergency Department patients. The second aim is to determine the impact of POC-guided decolonisation as compared to conventional laboratory testing on in-hospital infection rates with MSSA/MRSA in a pre-post-comparison study.

DETAILED DESCRIPTION:
The study EPICS-6 consists of three study phases. In phase one the novel POC-PCR-testing method for MSSA/MRSA-proof (cobas®LIAT®-System, Roche Molecular Systems Inc.) is technically established and integrated in Emergency Department procedures. After evaluation of processes and sample handling the second phase of this study assesses the prevalence of positive MSSA/MRSA-POC-testing in the general ED-population and in different risk groups. Based on the results of the previous study phases, the final phase comprises an interventional pre-post-comparison study. The interventional study assesses the impact of POC-result guided early decolonisation of MSSA/MRSA-colonized patients on in-hospital infection rates with MSSA/MRSA.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Emergency Department (ED) visit in one of the participating EDs

Exclusion Criteria:

* none

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
MSSA/MRSA prevalence in a general ED-population | on admission to the ED
  number of patients with a positive POC-test result for nasal/oral MSSA/MRSA
MSSA/MRSA in-hospital infection rates | at discharge from hospital for up to 90 days after admission
  number of in-hospital MSSA/MRSA infections in patients with known nasal/oral colonization with MSSA/MRSA. This outcome measure will be assessed for the time period between admission and discharge from hospital for up to 90 days after study inclusion. It will be assessed by routine MSSA/MRSA in-hospital testing and the respective test results will be retrieved from the hospital Information system.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin - Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No